CLINICAL TRIAL: NCT02158845
Title: Effects of the Levonorgestrel-releasing Intrauterine System Compared With the Leuprolide Acetate in Patients With Endometriosis: a Randomized Trial
Brief Title: Levonorgestrel-releasing Intrauterine System in Patients With Endometriosis
Acronym: SIU-LNG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Carolina Sales Vieira, Medical Doctor, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SIU-LNG 001
Record Dates: First submitted 2014-05-31; First posted 2014-06-09 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Endometriosis
Keywords: endometriosis; blood coagulation; levonorgestrel; GnRH agonist; progesterone-releasing intrauterine device
MeSH Terms: conditions — Endometriosis; Thrombosis | interventions — Levonorgestrel; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LNG-IUS (Active Comparator): LNG-IUS: levonorgestrel intrauterine system
  Interventions: Drug: LNG-IUS: levonorgestrel intrauterine system
- GnRHa (Active Comparator): GnRHa: leuprolide
  Interventions: Drug: GnRHa: leuprolide

INTERVENTIONS:
Drug: LNG-IUS: levonorgestrel intrauterine system — LNG-IUS (levonorgestrel intrauterine system) is inserted until the fifth day of the cycle. It releases 20 mcg/day of LNG
  Other Names: Mirena
  Arms: LNG-IUS
Drug: GnRHa: leuprolide — 3.75 mg leuprolide injected intramuscularly on a monthly basis
  Other Names: Lupron
  Arms: GnRHa

SUMMARY:
The hemostatic and inflammatory systems may activate each other. Endometriosis is a chronic inflammatory disease affecting 10% of women. The objective of this study is to compare the hemostatic effects of two treatments widely prescribed to women with endometriosis: the levonorgestrel intrauterine system (LNG-IUS) and the gonadotropin-releasing hormone analog (GnRHa) leuprolide acetate.

Hypothesis:

H0: There is no alteration in hemostatic system with the use of GnRHa or LNG-IUS H1: There is alteration in hemostatic system with the use of GnRHa or LNG-IUS

DETAILED DESCRIPTION:
Materials and Methods: In this randomized open-label controlled trial, 44 women with endometriosis will be randomly allocated to one of two groups: 22 women will be assigned to use LNG-IUS and 22 to use GnRHa. The assessed variables will be D-dimers, fibrinogen, prothrombin time, activated partial thromboplastin time, coagulation factors (F) II, V, VII, VIII, IX, X, and XI, antithrombin (AT), protein C, free protein S, tissue plasminogen activator (t-PA), α2-antiplasmin, thrombin-antithrombin complex, and prothrombin fragment 1+2. All variables will be assessed before treatment and six months after treatment onset.

ELIGIBILITY:
Inclusion Criteria:

* to have endometriosis
* aged 18 to 40 years
* Being without contraceptives for at least 3 months or with depot medroxyprogesterone acetate or GnRHa for at least 6 months at the time of randomization.

Exclusion Criteria:

* obese patients with a body mass index (BMI) ≥30 kg/m2
* smokers
* diabetics
* alcohol or drug users
* patients currently wishing to conceive
* patients with chronic diseases (except endometriosis)
* patients with infectious processes
* patients with a personal and/or family history of thromboembolic events
* patients taking medications known to interfere with inflammation markers (such as hormonal and nonhormonal anti-inflammatory agents) within the 15 days before the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
change from baseline in d-dimer | baseline and 6 months
  to compare the change over 6 months (6 months - baseline) on d-dimer of two treatments widely prescribed to women with endometriosis, LNG-IUS and GnRHa leuprolide acetate.

SECONDARY OUTCOMES:
change from baseline in Coagulation times | baseline and 6 months
  To compare the change over 6 months (6 months - baseline) of coagulation times as a composite measure of 3 variables: Thrombin time (TT), activated partial thromboplastin time (APTT), and prothrombin time (PT)
change from baseline in procoagulatory variables | baseline and 6 months
  to compare the change over 6 months (6 months - baseline) on procoagulatory variables (Fibrinogen, coagulation factors II, V, VII, VIII, IX, X, and XI) of two treatments widely prescribed to women with endometriosis, LNG-IUS and GnRHa leuprolide acetate.
Change from baseline in natural anticoagulants | baseline and 6 months
  to compare the change over 6 months (6 months - baseline) on natural anticoagulants (Protein C and antithrombin) of two treatments widely prescribed to women with endometriosis, LNG-IUS and GnRHa leuprolide acetate.
Change in activation of the coagulation cascade markers | baseline and 6 months
  to compare the change over 6 months (6 months - baseline) on activation of the coagulation cascade markers (concentrations of the thrombin-antithrombin complex and prothrombin fragment 1+2) of two treatments widely prescribed to women with endometriosis, LNG-IUS and GnRHa leuprolide acetate.
Change from baseline on antifibrinolytic variables | Baseline and 6 months
  to compare the change over 6 months (6 months - baseline) on antifibrinolytic variables (Plasminogen activator inhibitor 1, α-2 antiplasmin) of two treatments widely prescribed to women with endometriosis, LNG-IUS and GnRHa leuprolide acetate.

CONTACTS AND LOCATIONS:
Overall Officials: CAROLINA S VIEIRA, MD, PhD, Principal Investigator — Sao Paulo University
Locations (1):
- Hospital das Clinica de Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] Yamaguti EM, Brito MB, Ferriani RA, Garcia AA, Rosa-e-Silva JC, Vieira CS. Comparison of the hemostatic effects of a levonorgestrel-releasing intrauterine system and leuprolide acetate in women with endometriosis: a randomized clinical trial. Thromb Res. 2014 Dec;134(6):1193-7. doi: 10.1016/j.thromres.2014.09.014. Epub 2014 Sep 20. PMID 25283586